CLINICAL TRIAL: NCT00195780
Title: An Open-Label Study to Evaluate the Safety of Depakote ER in the Treatment of Mania Associated With Bipolar I Disorder in Children and Adolescents
Brief Title: A Study for the Treatment of Mania Associated With Bipolar I Disorder in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03-647
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Depakote
MeSH Terms: interventions — Valproic Acid

INTERVENTIONS:
Drug: Divalproex Sodium (Depakote ER)

SUMMARY:
The purpose of the study is to evaluate the long-term safety profile of the Investigational Medication Depakote ER in the treatment of Bipolar I Disorder, manic or mixed episode, in children and adolescents ages 10-17.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 10 and 17 years of age, inclusive, on Day 1 and weighs at least 60 lbs (27 kg).
* Subject has a current psychiatric diagnosis of bipolar I disorder, manic or mixed episode, based on the K-SAD-PL interview and DSM-IV-TR criteria.
* Subject is an outpatient in a manic or mixed episode with a YMRS score of greater than or equal to 16 during Screening and at Day 1.

Exclusion Criteria:

* Has an Axis I disorder other than Attention Deficit Hyperactivity Disorder (ADHD), Obsessive Compulsive Disorder (OCD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), Panic Disorder, Enuresis, Encopresis, Parasomnias, Agoraphobia, Specific Phobia, Social Phobia or Separation Anxiety Disorder; or subject has an Axis II disorder that would interfere with the subject's ability to comply with study procedures or confound interpretation of the study results. Subject meets DSM-IV-TR criteria for substance abuse within the month prior to Screening, or meets the criteria for substance dependence within the three months prior to Screening, or exhibits signs of drug or alcohol intoxication or withdrawal at Day 1.
* Is expected to require hospitalization for the current manic or mixed episode.
* Is violent, homicidal, or suicidal such that, in the opinion of the investigator, the subject is at significant imminent risk of hurting self or others.
* Has a history of a chronic or acute medical disorder that, in the opinion of the investigator, would preclude compliance with the protocol, or confound interpretation of the study results.
* Has a history of, or is suspected of having a seizure disorder.
* Has any central nervous system (CNS) neoplasm, CNS infection, demyelinating disease, degenerative neurological disease, or any progressive CNS disease.
* Has Platelet count less than or equal to 100,000/µL
* Has blood chemistry ALT/AST value(s) greater than or equal to 2 times upper limit of normal at screening.
* Is taking a protocol allowed medication for ADHD that has not been stable for at least 3 months prior to Day 1, or that, in the investigator's opinion, may be exacerbating mood symptoms.
* Requires anticoagulant drug therapy.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2005-02

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Y-MRS
CGI-S
C-GAS
CDRS-R
CGSQ
responders
remitters

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (29):
- United States (29):
  - PCSD Feighner Research, San Diego, California
  - PCSD Feighner Research, San Marcos, California
  - Altamonte Springs, Florida
  - Segal Institute for Clinical Research, Fort Lauderdale, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Kolin Research Group, Winter Park, Florida
  - Northlake Medical Research Center, Decatur, Georgia
  - Mountain West Clinical Trials, Eagle, Idaho
  - Capstone Clinical Research, Libertyville, Illinois
  - Clinco, Terre Haute, Indiana
  - Cientifica Inc., Newton, Kansas
  - Psychiatric Associates, Overland Park, Kansas
  - Brentwood Research Institute, Shreveport, Louisiana
  - Acadia Hospital, Bangor, Maine
  - Pharmasite Research, Baltimore, Maryland
  - North Carolina Neuropsychiatry, PA, Chapel Hill, North Carolina
  - Odyssey Research, Fargo, North Dakota
  - Neuro Behavioral Clinical Research, INC., Canton, Ohio
  - Psychiatric Professional Services, Cincinnati, Ohio
  - Rakesh Ranjan, M.D. & Associates, Inc., Lyndhurst, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Clinical Trials Specialists, Bala-Cynwyd, Pennsylvania
  - UTHSC, Sept. of Psychiatry, College of Medicine, Memphis, Tennessee
  - InSite Clinical Research, DeSoto, Texas
  - Red Oak Psychiatry, Houston, Texas
  - R/D Clinical Research, Lake Jackson, Texas
  - Northwest Clinical Research Center, Bellevue, Washington